CLINICAL TRIAL: NCT03942614
Title: Nordic Pole Walking for Individuals With Cancer: A Feasibility Study Assessing Physical Function and Health-Related Quality of Life
Brief Title: Nordic Pole Walking for Individuals With Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ontario Institute of Technology (Other)
Collaborators: Lakeridge Health Corporation (Other); Southlake Regional Health Centre (Other)
Responsible Party: Principal Investigator, Mika Nonoyama, Assistant Professor, University of Ontario Institute of Technology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 15-018
Record Dates: First submitted 2019-04-26; First posted 2019-05-08 (Actual); Last update posted 2019-05-08 (Actual); Status verified 2019-05

CONDITIONS: Cancer; Neoplasms
Keywords: Nordic Pole Walking; Exercise; Rehabilitation
MeSH Terms: conditions — Neoplasms; Motor Activity | interventions — Nordic Walking

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nordic pole walking (Experimental): walking with a pair of poles customized to an individual's height and stride length
  Interventions: Behavioral: Nordic pole walking
- Control (No Intervention): usual daily routine and activities of daily living

INTERVENTIONS:
Behavioral: Nordic pole walking
  Arms: Nordic pole walking

SUMMARY:
Individuals diagnosed with cancer tend to be inactive and have symptom burdens that impact quality of life. A community-based Nordic Pole Walking (NPW) program may help. The primary objective of this study was to see if it was feasible to do to a larger trial. The secondary objective was to determine the effects of NPW on physical function and health-related quality of life (HRQoL). NPW or no NPW was randomly assigned to adults with non-small cell lung, prostate, colorectal, and endometrial. Eight people were enrolled in the study with 4 in the NPW group (1 dropped out) and 4 in the no NPW group.

DETAILED DESCRIPTION:
Individuals diagnosed with cancer tend to be inactive and have symptom burdens that impact quality of life. An individualized, community-based Nordic pole walking (NPW) program may help. The primary objective of this study was to assess feasibility using the Thabane Framework of a randomized controlled trial (RCT). The secondary objective was to determine the effects of NPW on physical function (six-minute walk test, 30-second [30-s] chair stand test, Unsupported Upper Limb Exercise Test, handgrip strength, physical activity [PA]), and health-related quality of life (HRQoL, 36-Item Short Form Health [SF-36]). The study design was an eight-week multi-centred block randomized controlled feasibility study (no blinding) comparing a NPW program (versus usual daily routine) for adults with non-small cell lung, prostate, colorectal, and endometrial cancer, from hospitals and cancer support groups.

ELIGIBILITY:
Inclusion Criteria:

* a primary diagnosis (including reoccurrence) of histologically confirmed stage I-IV NSCLC, prostate, colorectal, or endometrial cancer (with any concurrent cancer treatment)
* a cancer diagnosis or treatment within the last three years
* ≥ 55 years old
* approval by the primary treating physician
* ability to communicate in English.

Exclusion Criteria:

• engaged in NPW within the last six-months

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2015-12-16 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Feasibility (assessed by qualitative field notes) | 8 weeks
  Feasibility was assessed using the framework as described by: Thabane L et al (2010) A tutorial on pilot studies: the what, why and how. BMC Medical Research Methodology, vol 10. England, p 1.
  The Thabane Framework uses 4 criteria to measure feasibility: Process, Resources, Management and Scientific. For each criteria, detailed field notes regarding objectives and measures were maintained throughout the study. These notes on the four Thabane criteria were used to categorize the study to one of four possible outcomes: 1) stop - the study is not feasible; 2) continue, but modify the protocol - the study is feasible with modifications; 3) continue without modifications, but monitor closely - the study is feasible with close monitoring; and 4) continue without modifications - the study is feasible as is.

SECONDARY OUTCOMES:
6-minute walk test (6MWT) | 8 weeks
  The 6MWT is a measure of submaximal functional capacity. Average healthy norms (61 to 80 years old) range from 583m (women) to 687m (men).
30-second chair stand test | 8 weeks
  The 30-s chair stand test is a measure of lower body strength. In 60 to 94 years olds, average healthy norms range from 13 (women) to 14 (men)
Unsupported Upper Limb Exercise Test (UULEX) | 8 weeks
  UULEX, an incremental test that measures peak unsupported arm exercise capacity. UULEX average healthy norms (40 to 89 years old) range from 11 (women) to 12 minutes (men).
Hand grip strength | 8 weeks
  average healthy norms (60 to 79 years old) ranging from 24kg (women) and 41kg
Functional Assessment of Cancer Therapy-Lung (FACT-L) | 8 weeks
  The FACT-L is a measure of health-related quality of life and includes 4 general and 1 lung cancer symptom-specific domain. The general domains (27 questions) include: physical well-being (PWB), social/family well-being (SWB), emotional well-being (EWB), and functional well-being (FWB). The lung cancer symptom specific (LCS) domain (7 questions) evaluates symptoms that are commonly experienced by lung cancer patients (i.e. shortness of breath, weight loss, and chest tightness). Domain scores are then combined to calculate the Total Outcome Index (TOI) (TOI = PWB + FWB + LCS), Functional Assessment of Cancer Therapy - General (FACT-G) score (FACT G = PWB + SWB + EWB + FWB), and FACT-L score (FACT-L = FACT- G + LCS). TOI range 0 to 135 with higher score better quality of life.
36-Item Short Form Health (SF-36) Questionnaire | 8 weeks
  The SF-36 is a measure of generic health-related quality of life. It assesses 8 health concepts (scales): 1) limitations in physical activities because of health problems; 2) limitations in social activities because of physical or emotional problems; 3) limitations in usual role activities because of physical health problems; 4) bodily pain; 5) general mental health; 6) limitations in usual role activities because of emotional problems; 7) vitality; and 8) general health perceptions. Scoring is a two-step process. First, precoded numeric values are recoded per a scoring key. In addition, each item is scored on a 0 to 100 range so that the lowest and highest possible scores (quality of life) are 0 and 100, respectively. Scores represent the percentage of total possible score achieved. In step 2, items in the same scale are averaged together to create the 8 scale scores. More information: https://www.rand.org/health-care/surveys_tools/mos/36-item-short-form/scoring.html.
International Physical Activity Questionnaire (IPAQ) | 8 weeks
  The IPAQ is a measure physical activity level. Questions ask about walking, moderate-intensity activities, vigorous-intensity activities, and sitting during the following 4 domains: a) leisure time physical activity; b) domestic and gardening activities; c) work-related physical activity; and d) transport-related physical activity. Two types of scoring were done: 1) in categories (low activity levels, moderate activity levels or high activity levels), and 2) as a continuous variable (MET minutes a week). MET minutes represent the amount of energy expended carrying out physical activity and is a multiple of a person's estimated resting energy expenditure. One MET is what is expended when at rest. To get MET minutes a week from the IPAQ walking was considered 3.3 METS, moderate physical activity to be 4 METS and vigorous physical activity 8 METS. (reference: https://ugc.futurelearn.com/uploads/files/bc/c5/bcc53b14-ec1e-4d90-88e3-1568682f32ae/IPAQ_PDF.pdf)

OTHER OUTCOMES:
Demographic information | baseline
  A data collection form was used to collect demographic information including cancer diagnosis and treatments, side effects, general health history, and smoking status (baseline only). No formal scale was used to collect this information; only descriptive information was collected.
Resting heart rate | baseline and 8 weeks
  beats per minute
Oxygen saturation | baseline and 8 weeks
  in %
Height | baseline and 8 weeks
  meters
Weight | baseline and 8 weeks
  meters
Body mass index | baseline and 8 weeks
  calculated as height divided by weight squared
Bicep circumferences | baseline and 8 weeks
  cm
Chest circumference | baseline and 8 weeks
  cm
Waist circumference | baseline and 8 weeks
  cm
Hip circumference | baseline and 8 weeks
  cm
Thigh circumferences | baseline and 8 weeks
  cm

IPD SHARING:
Plan to Share IPD: No
Sharing upon request.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-10-02): https://cdn.clinicaltrials.gov/large-docs/14/NCT03942614/Prot_SAP_000.pdf